CLINICAL TRIAL: NCT06939465
Title: Esophageal Visceral Hypersensitivity and Hypervigilance in Disorders of Gut-brain Interaction: the Roles of Cognitive-behavioral Therapy
Brief Title: Cognitive-behavioral Therapy for the Diseases Associated With Esophageal-brain-gut Axis Communication Abnormalities.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hualien Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Lei, Wei-Yi, Gastroenterology attending physician, Hualien Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCRD113-042
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Gut-Brain Disorders; GERD Without Erosive Esophagitis
Keywords: gastroesophageal reflux disease; disorders of gut-brain interaction; cognitive behavior therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral therapy (CBT) (Active Comparator): Cognitive Behavioral Therapy (CBT) will be implemented according to the following steps: (1) Psychoeducation and beginning of tracking; (2) Introduction to heart rate variability and breathing; (3) Cognitive restructuring and breathing application; (4) Cognitive defusion and behavioral experiments; (5) Coping strategies for problem-focused and emotion-focused approaches; (6) Conclusion of therapy and relapse prevention.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Lifestyle management (sham control) (Sham Comparator): Lifestyle management (sham control) will be implemented according to the following steps: (1) Psychoeducation and beginning of tracking; (2) Dietary habits: What, when, where, and why; (3) Changing my diet: Strategies and barriers; (4) Lifestyle factors: Alcohol, smoking, and sugar; (5) Lifestyle factors: Sleep and exercise; (6) Conclusion of therapy and relapse prevention.
  Interventions: Behavioral: Lifestyle management (sham control)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The participants will undergo a 6-week cognitive behavioral therapy (CBT) guided by a psychologist, with one session per week, each lasting 1 hour.
  Arms: Cognitive behavioral therapy (CBT)
Behavioral: Lifestyle management (sham control) — The participants will undergo a 6-week lifestyle management (sham control) guided by a psychologist, with one session per week, each lasting 1 hour.
  Arms: Lifestyle management (sham control)

SUMMARY:
Gastroesophageal reflux disease (GERD) is a challenging gastrointestinal disorder, and proton pump inhibitors (PPIs) are typically the first line of treatment. However, up to 40% of GERD patients experience little to no relief or only partial relief of their symptoms after receiving PPI therapy. Among these patients, who do not respond to high-dose PPIs taken twice daily, more than 90% exhibit conditions related to brain-gut axis communication disorders, such as esophageal hypersensitivity and functional heartburn. Visceral hypersensitivity and esophageal hypervigilance are the two key causes of esophageal symptoms in this group of patients. According to the Rome IV consensus on esophageal disorders, five categories are identified: functional chest pain, functional heartburn, globus sensation, functional dysphagia, and esophageal hypersensitivity. The diagnostic criteria state that patients must have chronic esophageal symptoms, and any structural, inflammatory, or motility abnormalities must be excluded. Therefore, diagnosing brain-gut axis communication disorders in the esophagus requires upper gastrointestinal endoscopy, esophageal pH-impedance testing, and high-resolution esophageal manometry. Neuromodulators, which regulate peripheral and central pain sensitivity, are a cornerstone of pharmacological treatment for brain-gut axis communication disorders and associated symptoms. Additionally, growing evidence supports the use of brain-gut axis behavioral therapies, such as gut-directed hypnotherapy and cognitive behavioral therapy (CBT), to effectively treat these disorders. However, research on neuromodulators and CBT in brain-gut axis communication disorders remains limited, and their efficacy is still unclear. The aim of this study is to investigate the effectiveness and role of CBT in treating brain-gut axis communication disorders. The information gained from this research will help clarify the pathophysiological mechanisms related to brain-gut axis communication abnormalities and refractory GERD symptoms. Furthermore, the findings will guide the development of effective treatment strategies for patients with brain-gut axis communication disorders who do not respond to PPI therapy in clinical practice.

DETAILED DESCRIPTION:
All participants will undergo questionnaire assessments and heart rate variability (HRV) measurements prior to treatment. The questionnaires include the Gastroesophageal Reflux Disease Questionnaire (GERDQ), PROMIS GERD, DSI & GSS, RSI, the Brief Esophageal Dysphagia Questionnaire (BEDQ), the Esophageal Hypersensitivity and Anxiety Scale (EHAS), Visceral Sensitivity Index (VSI), Sleep and Psychosocial Questionnaires (Pittsburgh Sleep Quality Index [PSQI], Taiwan Depression Questionnaire [TDQ], State-Trait Anxiety Inventory [STAI], Functional Dyspepsia [FD] Questionnaire, Irritable Bowel Syndrome [IBS] Questionnaire, and Quality of Life Questionnaire [SF-12, Northwestern Esophageal Quality of Life Questionnaire NEQOL]). HRV measurements will be conducted using a non-invasive "MindTech" physiological feedback system (Ministry of Health and Welfare Medical Device License No. 011374).

Afterwards, a single-blind trial with computer-generated random allocation will be conducted. Participants will undergo either six weeks of cognitive behavioral therapy (CBT) led by a therapist or six weeks of lifestyle management (sham control). Each group will receive one session per week, with each session lasting one hour. After six weeks of counseling, participants will undergo another round of questionnaire assessments and HRV measurements at the 12th week of the study. The questionnaire assessment and HRV measurements will take approximately 20 to 30 minutes to complete.

Cognitive behavioral therapy (CBT) will follow these steps in sequence: (1) education and tracking initiation, (2) introduction to heart rate variability and breathing, (3) cognitive restructuring and breathing techniques, (4) cognitive diffusion and behavioral experiments, (5) problem-focused and emotion-focused coping strategies, (6) conclusion of therapy and relapse prevention.

Lifestyle management (sham control) will follow these steps in sequence: (1) education and tracking initiation, (2) dietary habits: what, when, where, why, (3) changing my diet: strategies and obstacles, (4) lifestyle factors: alcohol, smoking, and sugar, (5) lifestyle factors: sleep and exercise, (6) conclusion of therapy and relapse prevention.

In this study, we will use a non-invasive physiological signal sensor connected to the physiological feedback system to measure participants' physiological signals, including electrocardiogram (ECG) and respiration. Prior to measurement, participants will be attached with ECG electrodes for a two-lead ECG, which will be converted into heart rate variability indicators. Additionally, a non-invasive respiratory sensor will measure the participant's breaths per minute. Except for a very small percentage of participants who may experience allergic reactions to ECG electrodes, the likelihood of adverse effects is less than 1%.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, with clear consciousness and willingness to sign the informed consent form.
2. Subjects with chronic esophageal symptoms related to disorders of the brain-gut axis communication (such as heartburn, acid reflux, sensation of a foreign body in the throat, difficulty swallowing, and chest pain or discomfort).

Exclusion Criteria:

1. Esophageal strictures, or history of surgery on the esophagus, gastrointestinal tract, or throat.
2. Structural esophageal diseases (such as diverticula, esophageal rings, etc.), infectious esophagitis, erosive esophagitis, eosinophilic esophagitis.
3. Non-erosive gastroesophageal reflux disease or significant esophageal motility disorders.
4. History of or current diagnosis of malignancies in the esophagus, gastrointestinal tract, or other organs.
5. Significant endocrine or rheumatic immune diseases that may affect gastrointestinal motility.
6. Continuous use of medications that may affect esophageal motility within the past month (such as anticholinergics, opioid-like agents, nitrates, calcium channel blockers, etc.).
7. Use of or currently taking antidepressants, selective serotonin reuptake inhibitors, or other psychotropic medications within the past three months.
8. Pregnant or breastfeeding women.
9. Individuals with mental illness or those who are unable to cooperate.
10. Known allergy to tricyclic antidepressants.
11. Known allergy to selective serotonin reuptake inhibitors.
12. Known allergy to any component of proton pump inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastroesophageal Reflux Disease Questionnaire（GERDQ） | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The minimum score of the questionnaire is 0 and the maximum score is 18. The higher the score, the worse the gastroesophageal reflux symptoms.
PROMIS Gastroesophageal Reflux Disease Questionnaire（PROMIS GERD） | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The minimum score of the questionnaire is 0 and the maximum score is 52. The higher the score, the worse the gastroesophageal reflux symptoms.
Disease symptom index(DSI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The minimum score of the questionnaire is 0 and the maximum score is 16. The higher the score, the worse the gastroesophageal reflux symptoms.
Reflux Symptom Index(RSI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The minimum score of the questionnaire is 0 and the maximum score is 45. The higher the score, the worse the gastroesophageal reflux symptoms.
The Brief Esophageal Dysphagia Questionnaire(BEDQ) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The lowest score of the questionnaire is 0 and the highest score is 40. The higher the score, the more severe the dysphagia.
Esophageal Hypervigilance and Anxiety Scale(EHAS) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The lowest score of the questionnaire is 0 and the highest score is 60. The higher the score, the more severe the esophageal hypervigilance and anxiety.
Visceral sensitivity index(VSI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The lowest score of the questionnaire is 0 and the highest score is 75. The higher the score, the higher the visceral sensitivity.
Pittsburgh Sleep Quality Index(PSQI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The lowest score of the questionnaire is 0 and the highest score is 21. The higher the score, the worse the sleep quality.
Taiwanese Depression Questionnaire(TDQ) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The lowest score of the questionnaire is 0 and the highest score is 54. The higher the score, the higher the depression index.
The State-Trait Anxiety Inventory(STAI) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The lowest score of the questionnaire is 1 and the highest score is 80. The higher the score, the more obvious the anxiety trait.
Illness Cognition Questionnaire (ICQ) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The lowest score of the questionnaire is 1 and the highest score is 72. The higher the score, the higher the level of disease awareness.
Short-form-12-health-survey-questionnaire(SF-12) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The results of the SF-12 health scale mainly include two total scores: physical health total score (PCS) and mental health total score (MCS). These two scores are used to measure an individual's health status in these two aspects.
  1. **Physical Health Score (PCS) and Mental Health Score (MCS)** are usually expressed as standardized scores with a mean of 50 and a standard deviation of 10.
  2. A higher score indicates better health, whereas a lower score indicates worse health.
Northwest Esophageal Quality of Life Scale(NEQOL) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The lowest score of the questionnaire is 0 and the highest score is 56. The higher the score, the worse the esophageal quality of life.
Global Symptom Severity Questionnaire(GSS) | Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  Each participant will undergo a questionnaire assessment upon entering the study, and another questionnaire assessment will be conducted at the end of the 12-week treatment period.
  The minimum score of the questionnaire is 0 and the maximum score is 100. The higher the score, the worse the gastroesophageal reflux symptoms.
Heart rate variability(HRV) | Participants will undergo heart rate variability measurement before receiving treatment, and another heart rate variability measurement will be conducted after week 12 of the study.
  Participants will undergo heart rate variability measurement before receiving treatment, and another heart rate variability measurement will be conducted after week 12 of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital,Buddhist Tzu Chi Medical Foundation, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT06939465/Prot_000.pdf
  • Informed Consent Form (2024-11-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT06939465/ICF_001.pdf